CLINICAL TRIAL: NCT00292578
Title: NAET® Testing Devices in Detection of Hypersensitivity to Cane Sugar
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nambudripad's Allergy Research Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Hypersensitivity to Cane Sugar; narfoundation 112
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Allergy; Fatigue; Hypoglycemia; Hyperglycemia; Indigestion
Keywords: Allergy; Sugar Intolerance; Fatigue
MeSH Terms: conditions — Hypersensitivity; Fatigue; Hypoglycemia; Hyperglycemia; Dyspepsia

INTERVENTIONS:
Procedure: NAET Testing Modalities

SUMMARY:
Background: Studies have noted a correlation between food sensitivities and health disorders. Various commonly seen health problems may be caused by cane sugar since it is lavishly and frequently used by people worldwide.

Objective: This study evaluated the efficacy of NAET testing instruments in detecting hypersensitivities to cane sugar.

Materials and Methods: Seventy-four subjects volunteered for this study. They were asked to write down one of their major health problems, the amount of sugar consumed on a daily basis and any known health problem(s) related to sugar consumption. The following testing modalities were used in the study: (1). Allergy Symptom-Rating Scale (ASRS); (2). NST Rating Scale (NSTRS); (3). Pulse Difference Rating Scale (PDRS). Test-1 was done twice. Tests 2 and 3 were done three times each: once without contacting sugar and then contacting sugar at one minute and ten minutes.

DETAILED DESCRIPTION:
NAET® testing devices are able to detect various levels of sensitivities to food substances in people (JNECM Vol. 1, No.1 & 2, 2005) before they manifest in symptoms. Using NAET testing devices various levels of sensitivities to sugar can be easily detected and the people who are found to be sensitive to sugar can be advised to take strict preventive measures thus helping to alleviate their health problems.

Primary Objective of the Study The study will evaluate the efficacy of NAET® testing devices in detecting sensitivity to cane sugar (intolerance, hypersensitivity, or allergy) in a group of subjects from both sexes who had no prior knowledge of any health problems related to sugar consumption.

Sample Characteristics Eighty subjects from a group of medical professionals of both sexes who came to attend a medical conference volunteered to participate in the study. These volunteers came from different parts of Japan thus representing a large part of the country. Nine NAET® practitioners volunteered to supervise the entire study.

An on-site invitation to participate in the study was given to a group of 80 medical professionals who had come to attend a medical conference in Tokyo, Japan. The invitation to take part in the study was given to each member in the same morning at the time of registration for the conference. The 80 subjects who responded to the invitation were asked to complete an Allergy Symptom Rating Scale. They were asked to list an approximate amount of daily sugar consumption in number of teaspoons. They were also asked to record if they had suffered from any known sugar-related problems in the past. The five volunteer-subjects with known diabetes and hypoglycemia were excluded from the study.

All 75 subjects had completed the Allergy Symptom Rating Scale form (ASRS) initially prior to entering the study. After enrolling in the study, the examiners performed the Neuromuscular sensitivity testing (NST Rating Scale) on their subjects before touching the test sample and recording of the results. Initial radial pulse was taken and recorded.

(Detailed information on the Allergy Symptom-Rating scale (ASRS); NSTRS, and PDRS: Subject were asked to mark and rate their symptoms in their own words on a zero to ten scale where zero=normal; and ten=maximum discomfort): 0= no allergy; (1-3)=1=mild; (4-6)= 2=moderate; (7-10)=3=severe. After the initial testing (after completing ASRS form, NSTRS after balancing the body, and after initial pulse reading) each one of the subjects was given a test tube with clear liquid (dissolved sugar) in their hands. The examiners tested the NST of the subjects with them holding the sample-test tube in their hands and the results recorded. The radial pulse was also checked and recorded. Then they were asked to continue to hold the samples for full ten minutes. At the end of ten minutes, they were assigned to be tested for NST and Pulse by different examiners. While still holding the test tube in the hand, the radial pulse was tested and recorded; NST was perfomed and recorded and each one of them was asked to complete another Allergy Symptom Rating Scale.

After completing the initial test, the monitors moved the subjects one at a time to a different area and each one of them was asked to continue to hold the sample-tubes in their hands for the following ten minutes.

At the end of ten minutes' waiting period with the test tubes in their hands, each subject was given another ASRS form to record their symptoms one more time. They were also instructed to rate their symptoms on a zero to ten scale. Then the monitors ushered them to different examiners to check the NST and radial pulse one more time, while still holding the test tubes in their hands. The results were recorded in a separate paper and the monitors collected the results and sent for analysis.

ELIGIBILITY:
Inclusion Criteria:

Allergy to foods Undiagnosed health problems -

Exclusion Criteria:

Cancer History of previous Anaphylaxis Any debilitating health problems

-

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-01; Study Completion 2006-01

PRIMARY OUTCOMES:
The study will evaluate the efficacy of NAET® testing devices in detecting sensitivity to cane sugar (intolerance, hypersensitivity, or allergy) in a group of subjects from both sexes who had no prior knowledge of any health problems related to sugar

SECONDARY OUTCOMES:
Improve opportunity to get better dietary management and guidance for a better life-style. This may reduce or prevent the risk of sugar-related problems at a later age.

CONTACTS AND LOCATIONS:
Overall Officials: Devi S Nambudripad, DC,L.Ac,PhD, Principal Investigator — NAR Foundation
Locations (1):
- 6714-32 Beach Blvd.,, Buena Park, California, United States